CLINICAL TRIAL: NCT05155683
Title: Comparative Study of the Use of Phototherapy and Ultrasound to Reduce Localized Fat
Brief Title: Combination of Light and Ultrasound to Reduce Abdominal Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Christiane Pavani, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MMS
Record Dates: First submitted 2021-11-03; First posted 2021-12-13 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Subcutaneous Fat Disorder
Keywords: LLLT; Cavitation; Photobiomodulation
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: The abdomen of the participants will be cleaned by using a neutral cleansing soap. Each participant will receive safety glasses for eye protection, which will also contribute to blindness of the study. PBM will be applied when using abdominal straps as developed by Cosmedical (Mauá, São Paulo, Brazil). The abdomen strap will be covered with a sheet and that will also help with the blindness of the study. After randomization, the study population will be divided into four groups (n= 10 per group), which are: (1) Group A - PBM with infrared LED application + sham ultrasound + muscle electrostimulation; (2) Group B - LED sham PBM + ultrasound + muscle electrostimulation; (3) Group C - combined treatment (PBM + ultrasound) + muscle electrostimulation; (4) Group D - sham combined treatment + muscle electrostimulation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither the participants involved in the study, nor the outcomes assessor will be aware of the groups formed, as well as the treatments received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Photobiomodulation (Active Comparator): PBM with infrared LED application + sham ultrasound + muscle electrostimulation
  Interventions: Device: Photobiomodulation (PBM) with infrared LED; Device: Muscle electrostimulation
- low frequency ultrasound (Active Comparator): LED sham PBM + LOFU + muscle electrostimulation
  Interventions: Device: Low-frequency ultrasound (LOFU); Device: Muscle electrostimulation
- Combined treatment (PBM + LOFU) (Active Comparator): Combined treatment (PBM + LOFU) + muscle electrostimulation
  Interventions: Device: Photobiomodulation (PBM) with infrared LED; Device: Low-frequency ultrasound (LOFU); Device: Muscle electrostimulation
- Sham Treatment (Sham Comparator): Sham combined treatment + muscle electrostimulation
  Interventions: Device: Muscle electrostimulation

INTERVENTIONS:
Device: Photobiomodulation (PBM) with infrared LED — All participants will receive 30 minutes of PBM (or PBM sham), with an abdominal strap containing 4 LED clusters with 72 devices that emit 830 nm wavelength with 20 nm spectral width, in continuous operating mode, 5 mW average radiant power per LED, 71 mW/cm² power density at aperture, 20.4 cm² of total area irradiated, 71 mW/cm² of irradiance at target, exposure duration of 1800 seconds, 127.8 J/cm² of radiant exposure, 2.6 kJ of radiant energy, per contact application technique, twice a week for a month, totaling 8 sessions.
  Other Names: Low-level light therapy (LLLT)
  Arms: Combined treatment (PBM + LOFU); Photobiomodulation
Device: Low-frequency ultrasound (LOFU) — Subsequently the demarcation of the target area for LOFU treatment (Thoor DGM Electronica, Santo André, São Paulo, Brazil), the application of the neutral conductive gel will occur for the use of low-frequency ultrasound for 30 minutes, which will occur with 22 cm² effective radiating area (ERA) size, <8 BNR emission intensity, 40 kHz frequency, continuous mode, 60W, 100 cm² of total treated area, twice a week for a month, totaling 8 sessions.
  Arms: Combined treatment (PBM + LOFU); low frequency ultrasound
Device: Muscle electrostimulation — The session will end with 20 minutes of Russian Current (Tensor DGM Electronica, Santo André, São Paulo, Brazil), whose carrier frequency occurs in 2500 Hz, which will be adjusted according to the parameters described by Evangelista et al. (2003), which are: pulse frequency of 30 Hz; up/down ramp of 2 seconds each; support/rest time of 13 seconds each. The current intensity used will be the maximum supported by each participant and that is comfortable and sufficient to provide visible contraction. The treatment will consist of eight sessions that will occur twice a week, totaling a month of treatment.

SUMMARY:
Light and ultrasound can be interesting alternatives to reduce abdominal fat. Thus, the main objective of this study will be to evaluate the effects of these isolated techniques and their association in subcutaneous abdominal localized fat. These techniques will be used adding muscle electrostimulation in all groups. A total of 40 female participants will be recruited at the university outpatient, which will be distributed among four experimental groups: light + sham ultrasound + electrostimulation; light sham + ultrasound + electrostimulation; combined treatment (light + ultrasound) + electrostimulation; sham combined treatment + electrostimulation. The treatments will consist of eight sessions, twice a week for a month, being 90 minutes per session.

DETAILED DESCRIPTION:
The search for the ideal shape and the lifestyle that favours the increase of adipose depots are some factors responsible for the increasing demand for procedures to reduce localized fat. It has been shown that photobiomodulation (PBM) and low-frequency ultrasound (LOFU) can be interesting alternatives to treat this aesthetic dysfunction. However, there is no consensus about the best parameters for the application of these therapeutic resources. Thus, the main objective of this study will be to evaluate the effects of these isolated techniques and their association in subcutaneous abdominal localized fat.This will be a controlled, randomised, double-blind, single-centred clinical trial. Infrared light emitting diode - LED - (830±20 nm, 71 milliwatt per square centimeter mW/cm², 127.8 J/cm²), low-frequency ultrasound (30 kilohertz (kHz), 3 W/cm²) and combination of techniques will be used, adding muscle electrostimulation in all groups (2500 Hz, 30 bps, 50%). A total of 40 female participants will be recruited at the university outpatient, which will be distributed among four experimental groups that will compose the pilot study: PBM + sham ultrasound + electromyostimulation; PBM sham + LOFU + electromyostimulation; combined treatment (PBM + LOFU) + electromyostimulation; sham combined treatment + electromyostimulation. At each session, the participants will receive 30 minutes PBM with an abdominal strap, subsequent demarcation on the target area to be treated with LOFU for 30 minutes and completion with 20 minutes of electrically induced muscle contraction. The treatments will consist of eight sessions, twice a week for a month. The main outcome of this study will be abdominal skinfold reduction and the secondary variables will be including anthropometric data, local temperature, nutritional routine and physical activity data, quality of life, self-esteem, satisfaction grade with the treatment and visual changes.

ELIGIBILITY:
Inclusion Criteria:

* BMI of between 18.5 and 27.5 kg/m² (normotrophic or overweight body mass);
* Fitzpatrick phototype from I to IV;
* Who have fat located in the abdominal region characterized by abdominal skinfold higher than 20 mm;
* Who are sedentary of perform physical activity whose intensity is equal to or less than 450 METs/minutes/week (metabolic equivalents = METs);
* Who have stabilized weight, that is, who have not acquired or eliminated more than 2.5 kg in the 6 months preceding the screening;
* Absence of signs/symptoms of disease.

Exclusion Criteria:

* Women who have used drugs that alter body composition in the last 3 months prior to starting treatments; who use sensitizing agents, diuretics or are undergoing photodynamic therapy;
* Participants who are undergoing aesthetic treatments to reduce abdominal/waist circumferences; those who have been previously submitted to abdominoplasty or liposuction surgeries; those who are on a diet therapy monitoring to reduce their measurements; those who are using or have taken drugs or food supplements in last 90 days, in order to reduce their measurements and their weight, which may affect their lipid metabolism, appetite or nutrients absorption; those who have been submitted previously to oophorectomy; those with signs and/or symptoms of climacteric at the menopause; pregnant or lactating women or who are planning a pregnancy before the end of treatment participation.
* Participants who have abdominal hernia; osteoporosis; phlebitis and thrombophlebitis; autoimmune diseases; cardiovascular problems (hypertension, cardiac insufficiency, arrhythmia, thrombosis); metabolic dysfunctions (diabetes and thyroid disorders); hepatitis or other liver diseases (non-alcoholic fatty liver disease, cirrhosis); respiratory issues (asthma, chronic obstructive pulmonary disease); haematological disturbances (anaemia); renal; dermatological (reduced sensitivity); digestive disorders (gastritis, ulcers); neurological (dementia or schizophrenia), or who have cognitive impairment that may compromise the proper understanding of informed consent; who have already been affected by important inflammatory processes and/or who have a history of cancer;
* Participants who present tattoos and/or piercings in the region to be treated, who use intrauterine devices, pacemakers, or other electromagnetic implants, as well as joint prostheses.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Abdominal skinfold change | Before the start (Day 0), after the fourth session (Day 15) and after the treatments (Day 30).
  This outcome will be measured in millimeters (mm) by direct reading using adipometer (Sanny, American Medical do Brasil Ltda., São Bernardo do Campo, Brazil).

SECONDARY OUTCOMES:
Anthropometric data (body weight) | Day 0, Day 15 and Day 30.
  Body weight will be measured in kilograms (kg) using a calibrated digital scale.
Anthropometric data (height) | Day 0.
  Height will be measured in centimeters (cm) and will be collected using a standard stadiometer.
Anthropometric data (body mass index) | Day 0, Day 15 and Day 30.
  The body mass index (BMI) will be calculated from data obtained from the weight (in kilograms) and height (in centimeters) of each participant. The final value will be provided in kg/cm².
Anthropometric data (waist circumference) | Day 0, Day 15 (body weight, BMI, waist and hip circumferences, abdominal and suprailiac skinfold only), and Day 30.
  A properly trained researcher will measure the waist circumference in centimeters (cm), respecting the reference points according to the World Health Organisation (WHO).
Anthropometric data (hip circumference) | Day 0, Day 15 and Day 30.
  A properly trained researcher will measure the hip circumference in centimeters (cm), respecting the reference points according to the World Health Organisation (WHO).
Anthropometric data (waist/hip circumference ratio) | Day 0, Day 15 and Day 30.
  The waist/hip circumference ratio will be obtained by dividing the values obtained in centimeters in order to verify a possible change in the cardiovascular risk profile.
Anthropometric data (skinfold measures) | Day 0, Day 15 (abdominal and suprailiac skinfolds only), and Day 30.
  A properly trained researcher will realize the skinfolds evaluation that allows to assess the prediction of body fat based on subcutaneous fat and body density and these will be collected using an adipometer according to the methodology proposed by Pollock and Wilmore (1993) for the measurements referring to the seven skinfolds - tricipital, subscapular, bicipital, suprailiac, abdominal, thigh and leg (medial calf) locations, which will be obtained in millimeters (mm).
Local temperature | Day 0 and Day 30.
  Thermographic image will be captured using a Compact Thermal Camera (C2, FLIR Systems, Oregon, USA), which calculates the temperature of a given surface through the infrared emission and it will allow verify if there will be any change in local temperature after treatment.
Bioimpedance analysis (weight) | Day 0 and Day 30.
  The weight (in kilograms) will be obtained from bioimpedance analysis (Biodynamics Corp., Shoreline - WA, USA) that will allow estimation of body components in a non-invasive way. To obtain legitimate values, each participant will be instructed to drink an average of 2 litres of water and avoid the use of diuretic medication on the day before the exam, do not perform physical activity for at least 12 hours before the test, do not drink alcohol or drinks containing caffeine, not having a menstrual period and, on the day of the exam, fasting of at least 4 hours will be necessary.
Bioimpedance analysis (fat mass percentage) | Day 0 and Day 30.
  The fat mass percentage (%) will be obtained from bioimpedance analysis (Biodynamics Corp., Shoreline - WA, USA) that will allow estimation of body components in a non-invasive way. To obtain legitimate values, each participant will be instructed to drink an average of 2 litres of water and avoid the use of diuretic medication on the day before the exam, do not perform physical activity for at least 12 hours before the test, do not drink alcohol or drinks containing caffeine, not having a menstrual period and, on the day of the exam, fasting of at least 4 hours will be necessary.
Bioimpedance analysis (lean mass percentage) | Day 0 and Day 30.
  The lean mass percentage (%) will be obtained from bioimpedance analysis (Biodynamics Corp., Shoreline - WA, USA) that will allow estimation of body components in a non-invasive way. To obtain legitimate values, each participant will be instructed to drink an average of 2 litres of water and avoid the use of diuretic medication on the day before the exam, do not perform physical activity for at least 12 hours before the test, do not drink alcohol or drinks containing caffeine, not having a menstrual period and, on the day of the exam, fasting of at least 4 hours will be necessary.
Nutritional assessment | Day 0, during the study period (3 times per week) and Day 30.
  The nutritional routine will be documented as follows: the 24-hour food recall will be collected at the time of the initial evaluation (D0); during treatment, participants will have to fill their daily diet at least three times a week on a nutritional planner, which should contain all the food eaten on those chosen days; and after the end of treatment (D30) the participants will answer again the 24-hour food recall.
Physical activity assessment | Day 0, Day 15 and Day 30.
  The physical exercises performed by the participants during the study will be registered using the International Physical Activity Questionnaire (IPAQ), short version.
Quality of life scale | Day 0 and Day 30.
  The WHOQOL-BREF (Brief version of the World Helath Organization quality of life questionanaire) is the smaller version of the WHOQOL-100 quality of life questionnaire. WHOQOL-BREF consists of 26 questions, whose answers follow a Likert scale (from 1 to 5, the higher the score, better is the quality of life). This questionnaire has 2 questions that assess quality of life in general, being that the others make up 4 domains (physical, psychological, social relations and environment).
Self-esteem scale | Day 0 and Day 30.
  The body shape questionnaire (BSQ) has 34 questions and each question has six possible answers, as follows: 1) Never, 2) Rarely, 3) Sometimes, 4) Often, 5) Very often and 6) Always. Quantification of the level of concern in relation to self-image is done through a sum of responses. Result less than or equal to 110 points indicates there is no concern; greater than 110 and less than or equal to 138 points indicates a slight concern; greater than 138 and less than or equal to 167 points indicates moderate concern and if greater than 168 points indicates serious concern.
Visual change assessment | Day 0 and Day 30.
  Visual change assessment will be investigated from standardized photograph captures. Participants will be instructed to wear bathing or gym clothes and they will be positioned with their backs to a black background wall, at a distance of 0.7 m from it, on a paper template fixed to the ground, as suggested by Dias et al., (2017). Then, a professional trained for this purpose will be positioned at a distance of 1 m from the participant and will capture four records of her, these being in the anterior, posterior and lateral positions (90° to the right and to the left). Focal length, room lighting and recording mode will also be standardized.
Satisfaction degree with treatment | Day 30.
  The participants satisfaction grade with the treatment will be verified by means of a questionnaire containing seven multiple choice questions prepared by our research group based on data contained in the literature. The degree of discomfort during the treatment will be evaluated; if discomfort occurred, for how long did it persist; the degree of satisfaction in relation to the results achieved; the percentage degree of improvement of the complaint; whether the observed effects were below, within or above what was expected; whether she would do the treatment again; and how much would it indicate the treatment for someone close to it with the same complaint.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Sena, MSc, Study Chair — PhD student
Locations (1):
- Universidade Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be shared after 3 months after manuscript publication
Access Criteria: Researchers who provide a methodologically sound proposal.